CLINICAL TRIAL: NCT06875804
Title: Effects of Compressive Myofascial Release of the Vastus Lateralis on Lateral Patellar Tracking in Patients With Patellofemoral Pain Syndrome
Brief Title: Compressive Myofascial Release of the Vastus Lateralis on Lateral Patellar Tracking in Patellofemoral Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0149
Record Dates: First submitted 2025-03-10; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain Syndrome; Myofascial Release; Vastus Lateralis; Patellar Tracking; Knee joint; Pain; Range of motion
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Baseline physical therapy treatment (Active Comparator): baseline physical therapy treatment
  Interventions: Other: baseline physical therapy treatment
- Group B: Compressive myofascial release of vastus lateralis. (Experimental): baseline physical therapy treatment along with compressive myofascial release of vastus lateralis
  Interventions: Other: Compressive myofascial release of vastus lateralis.

INTERVENTIONS:
Other: baseline physical therapy treatment — Group A focuses on pain relief, muscle relaxation, and strengthening. Hot packs and TENS are applied to the lateral thigh and knee for 20 minutes to reduce pain and muscle tension. Hip strengthening exercises include side-lying hip abduction, clam-shells, prone hip extension, bridging, and lunges. Quadriceps exercises involve straight leg raises, prone terminal knee extension, and mini-squats. Each exercise is done in 2-3 sets of 10-15 repetitions, holding stretches for 5 seconds.
  Arms: Group A: Baseline physical therapy treatment
Other: Compressive myofascial release of vastus lateralis. — The experimental group receives an additional session of Compressive Myofascial Release (CMFR) for the Vastus Lateralis to address lateral patellar tracking in PFPS patients. The patient lies on their side, and the therapist identifies tight areas, applying firm pressure for 20-30 seconds. Deeper pressure is held for 30-60 seconds, followed by 1-2 minutes of cross-fiber friction. The session includes muscle shaking for 30 seconds and stretching the Vastus Lateralis by extending the hip and flexing the knee for 30-60 seconds, repeated 2-3 times. Patient response is documented for progress tracking.
  Arms: Group B: Compressive myofascial release of vastus lateralis.

SUMMARY:
Patellofemoral Pain Syndrome is a prevalent condition characterized by anterior knee pain, often exacerbated by activities such as squatting, running, and stair climbing. This condition is frequently associated with improper patellar tracking, particularly lateral displacement, which can be influenced by various factors including muscular imbalances and tightness. The vastus lateralis muscle, part of the quadriceps group, is often implicated in contributing to lateral patellar tracking due to its attachment and alignment. Compressive myofascial release (CMFR) is a therapeutic technique aimed at reducing muscle tightness and restoring optimal muscle function. This study will explore the effects compressive myofascial release on the vastus lateralis in improving patellar tracking in patients diagnosed with Patellofemoral Pain Syndrome.The methodology of this study involves a randomized controlled trial with a sample of patients diagnosed with Patellofemoral Pain Syndrome. Non-probability convenience sampling technique will be used and participants will be recruited in groups after randomization. Participants(n=26) will be divided into two groups: the intervention group (n=13) receiving compressive myofascial release on the vastus lateralis, and a control group receiving(n=13) a routine treatment. The intervention will be administered over a period of four weeks, with sessions occurring three times weekly. Patellar tracking will be assessed using q-angle analysis both pre- and post-intervention. Additionally, subjective measures of pain and functional ability will be evaluated using the Numeric pain rating scale (NPRS) and the Kujala Patellofemoral Score. Data analysis will focus on comparing the changes in lateral patellar displacement and patient-reported outcomes between the two groups to determine the efficacy of compressive myofascial release in correcting lateral patellar tracking and alleviating symptoms of Patellofemoral Pain Syndrome. SPSS version 25 will be used for data analysis

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is one of the most common health-related complaints in today's societies. PFPS refers to a syndrome that comprises of the following signs and symptoms: anterior knee pain, inflammation, imbalance and instability. About 50% of the non-specific knee pain is diagnosed as PFPS. PFPS frequently becomes chronic, and patients cannot do physical activity. Individuals with PFPS typically report pain that is either located in the peri-patellar or retro-patellar region during active movements involving knee movement.

Myofascial pain syndrome (MPS) has been attributed as the main cause and primary source of musculoskeletal pain in 30-85% of the patients attending physical therapy clinics. Myofascial pain syndrome often presents in the forms of pain, muscle spasm or TrP. TrP has been described as a hyperirritability spot located in a taut band of muscle; or a small pea or rope-like nodular or crepitant (crackling, grating) area within the muscle, which is painful to palpation or compression and refers pain, tenderness, or an autonomic response to a remote area. It is stated that "jump response" is elicited when pressure is applied to a Trp. TrP may result from mechanical overload, trauma, overuse, postural faults, or psychological stress. Based on their primary functions, muscles are categorized as "phasic" or "postural" muscles. In response to dysfunction or overuse, the phasic muscles tend to be inhibited or weakened; while the postural muscles tend to develop higher tone and ultimately shorten. A muscle imbalance between the dynamic and postural muscles may lead to MTP in the musculoskeletal system.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 20 to 40 years
* Male and female gender
* Diagnosed cases of Patellofemoral syndrome
* Participants with positive J sign and Clarke's test
* Pain provoked during knee loading physical activity, such as jumping, running, squatting, or going up or down stairs in last 3 months
* Presence of excessive lateral patellar tracking on axial view radiographs

Exclusion Criteria:

* History of knee surgery in the past year.
* Any contraindications to myofascial release therapy, such as active infections, open wounds.
* Presence of hip pathology or other knee conditions such as ligament tears, meniscal injuries, Osgood-Schlatter or Sinding-Larsen-Johanssen syndrome or jumpers knee
* Participants with a history of trauma or repetitive episodes of patellar subluxation or dislocation
* Use of intra-articular corticosteroid injections
* Presence of auto-immune disorder (spondylolisthesis, spondylitis, Rheumatoid arthritis etc.) other than knee OA or systemic conditions such as severe cardiovascular disease

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 4 weeks
  It is a standardized self-report device consisting of a horizontal line used to estimate the subjective level of pain intensity. It is a 10 points numerical scale, corresponding to the degree of pain.
Q angle | 4 weeks
  Quadriceps angle (Q-angle) has been used as a diagnostic measurement to assess factors which appear to increase the risk of the development of acute and/or chronic patellofemoral injury and pain in bipedal individuals. The Q-angle is the angle between the line of pull of the quadriceps (anterior superior iliac spine to mid-patella) and a line connecting the center of patella with tibial tuberosity. Normal Q-angle for males is 10-13 degrees and 15-17 degrees for females.
Goniometry | 4 weeks
  A goniometer is the most common instrument used to measure range of motion. If a patient has altered range of motion in a particular joint, the therapist can use a goniometer to assess what the range of motion is at the initial assessment, and then make sure the intervention is working by using the goniometer in subsequent sessions to assess the effectiveness of the intervention. Goniometric measurements should be performed with functional AROM and PROM. The typical documentation for the knee motion is: 10-0-135 degrees beginning with hyperextension, moving through neutral 0 and into flexion.
Kujala score | 4 weeks
  The "Kujala Score" is the eponymous name for the Anterior Knee Pain Scale (AKPS). It is a patient-reported outcome survey and diagnostic tool that aims to assess the severity of symptoms and physical limitations in patients with patellofemoral pain syndrome (PFPS). It was initially derived due to the diagnostic inconsistency among other tools that were used with PFPS patients. The Kujala Patellofemoral Scale is a valid and reliable questionnaire to evaluate functioning in patients with PFPS. The scores range from a maximum of 100 to a minimum of 0, with lower scores indicating greater pain and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Fatima, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Social Security Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torrente QM, Killingback A, Robertson C, Adds PJ. The Effect of Self-Myofascial Release on the Pennation Angle of the Vastus Medialis Oblique and the Vastus Lateralis in Athletic Male Individuals: An Ultrasound Investigation. Int J Sports Phys Ther. 2022 Jun 1;17(4):636-642. doi: 10.26603/001c.35591. eCollection 2022. PMID 35693863
- [Background] Stanek J, Sullivan T, Davis S. Comparison of Compressive Myofascial Release and the Graston Technique for Improving Ankle-Dorsiflexion Range of Motion. J Athl Train. 2018 Feb;53(2):160-167. doi: 10.4085/1062-6050-386-16. Epub 2018 Jan 26. PMID 29373060
- [Background] Zago J, Amatuzzi F, Rondinel T, Matheus JP. Osteopathic Manipulative Treatment Versus Exercise Program in Runners With Patellofemoral Pain Syndrome: A Randomized Controlled Trial. J Sport Rehabil. 2020 Dec 17;30(4):609-618. doi: 10.1123/jsr.2020-0108. PMID 33333491
- [Background] Halabchi F, Abolhasani M, Mirshahi M, Alizadeh Z. Patellofemoral pain in athletes: clinical perspectives. Open Access J Sports Med. 2017 Oct 9;8:189-203. doi: 10.2147/OAJSM.S127359. eCollection 2017. PMID 29070955
- [Background] Schoots EJ, Tak IJ, Veenstra BJ, Krebbers YM, Bax JG. Ultrasound characteristics of the lateral retinaculum in 10 patients with patellofemoral pain syndrome compared to healthy controls. J Bodyw Mov Ther. 2013 Oct;17(4):523-9. doi: 10.1016/j.jbmt.2013.03.005. Epub 2013 Apr 26. PMID 24139014